CLINICAL TRIAL: NCT05288946
Title: Effect of Segmental Control Program on Hamstring Peak Torque,Pain,Function and Range of Motion in Patients With Non-specific Low Back Pain
Brief Title: Effect of Segmental Control Program on Hamstring Peak Torque in Patients With Non-specific Low Back Pain
Acronym: NSLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p.t.REC/012/002673
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Chronic Low-back Pain
Keywords: segmental stabilization exercise; low back pain; peak torque
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: segmental stabilization exercises
Who Masked: Investigator, Outcomes Assessor
Masking Description: random generator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- local segmental control and closed kinetic chain (Experimental): the patients will receive local segmental control and closed kinetic chain three times a week for four weeks
  Interventions: Other: local segmental control and closed kinetic chain; Other: traditional therapy
- local segmental control and open kinetic chain (Experimental): the patients will receive local segmental control and open kinetic chain three times a week for four weeks
  Interventions: Other: local segmental control and open kinetic chain; Other: traditional therapy
- traditional therapy (Active Comparator): the patients will receive traditional therapy three times a week for four week
  Interventions: Other: traditional therapy

INTERVENTIONS:
Other: local segmental control and closed kinetic chain — the patients will receive Lumbar multifidus activation and Transversus abdominis activation then closed kinetic chain exercise in the form of Stand-up position on unstable surface, Closed chain lunge exercises, with the addition of hand weights, Bridge in prone position, Bridge in supine position, Lateral Bridge
  Arms: local segmental control and closed kinetic chain
Other: local segmental control and open kinetic chain — the patients will receive Lumbar multifidus activation and Transversus abdominis activation then open kinetic chain in the form of Lower limb abduction, Knee extension in a supine position on a roller, Open chain exercise of the upper limb after co-contraction of transversus abdominis and multifidus.
  Arms: local segmental control and open kinetic chain
Other: traditional therapy — the patients will receive exercise in the form of Sitting knee raise on gym ball to maintain stability in the presence of hip movement on a reduced base of support, abdominal slide to control action of the rectus abdominis while moving, Lying trunk curl with leg lift to strengthen upper and lower abdominals (figure 1-6), Basic superman to strengthen the spinal and hip extensors

SUMMARY:
The purpose of this study is to investigate the effect of segmental control exercises program on hamstring peak torque, pain, function, and ROM in patients with non-specific low back pain.

DETAILED DESCRIPTION:
Low back pain (LBP) is a significant health problem internationally characterized by various biophysical, psychological, and social dimensions affecting functioning, societal participation, and personal financial prosperity.The reported prevalence of LBP was high, especially for chronic non-specific low back pain, approximately 15.4%. of which chronic low back pain was about 2.5 times more prevalent in the working population compared to the non-working group. Recently, there has been a focus on lumbar stabilization exercises that prove to be effective and may be superior to general exercises for LBP management. The approach is aimed at improving the neuromuscular control, strength, and endurance of the active subsystem stabilizing the spine. Several groups of muscles are particularly targeted namely, the transverses abdominis and the multifidus muscles that are central to maintain spinal and trunk stability. But also other core muscles are involved. so this study will be conducted to investigate the effect of segmental stabilization exercise on low back pain. forty-five patients will be allocated to three groups. first experimental will receive segmental stabilization phase 1 and phase 2, second experimental will receive segmental stabilization phase 1 and 3, the third one is the control group and receives traditional treatment

ELIGIBILITY:
Inclusion Criteria:

1. The patients had NS LBP Patients with age from 20 to 40 years for both genders.
2. The lumbar region of back pain lasts for 4 weeks & more has not been diagnose as a specific disease or spinal abnormality.
3. Mild to moderate disability according to the Oswestry Disability Index (ODI) (up to 40%).
4. Shortening of hamstring.
5. The study populations must be willing to participate in the study.

Exclusion Criteria:

1. Neurological, systemic illness and infectious diseases such as rheumatologic diseases, tumor, cardiovascular disease.
2. Psychiatric/mental deficit
3. Patients who had a previous surgical history (within 6 months) were also excluded prior to the baseline assessment.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
peak torque | up to four weeks
  isokinetic will be used for measuring hamstring peak torque

SECONDARY OUTCOMES:
pain intensity | up to four weeks
  visual analogue scale will be used for assessment of pain intensity
disability | up to four weeks
  oswestry disability scale will be used for assessment of disability, Each patient was asked to answer by checking one box in each section for the statement which best applies to him. Then the marks had been counted and divided by 50 or 45.score ranging from 0 (no pain or disability) to 50 (severe pain and disability) . Then was multiplied by 100 for the percentage (score/ 50) x 100=% points. A score of 0% to 20% is minimal disability, 21%-40%: moderate disability, 41%-60%: severe disability, 61%-80%: crippled and 81%-100%: complete disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt